CLINICAL TRIAL: NCT00982930
Title: A Phase III Open-Label Extension Study to Assess the Safety and Efficacy of Tobramycin Inhalation Powder After Manufacturing Process Modifications (TIPnew) in Cystic Fibrosis (CF) Subjects Who Completed Participation in Study CTBM100C2303.
Brief Title: Open Label Extension to Bridging Study CTBM100C2303
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100C2303E1; 2008-004764-39 (EudraCT Number)
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Pseudomonas Aeruginosa; Cystic Fibrosis
Keywords: Tobramycin Inhalation Powder; Cystic fibrosis; Lung diseases; Anti-Bacterial Agents
MeSH Terms: conditions — Pseudomonas Infections; Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tobramycin Inhalation Powder (TIP) (Experimental): Participants received 112 mg (four 28 mg capsules) of TIP administered by the T-326 Inhaler, twice a day (b.i.d.), given in a cycle of 28 days on treatment followed by 28 days off treatment (one cycle = 56 days) for up to 3 cycles.
  Interventions: Drug: Tobramycin inhalation powder

INTERVENTIONS:
Drug: Tobramycin inhalation powder — Tobramycin inhalation powder, 112 mg (4 capsules of 28 mg), inhalation capsules, b.i.d.

SUMMARY:
This was an open-label, single arm (uncontrolled) study in participants suffering from cystic fibrosis, who had completed their study participation in CTBM100C2303 (all visits) and who were proven infected with Pseudomonas aeruginosa (P. aeruginosa) at enrollment into CTBM100C2303.

ELIGIBILITY:
Inclusion Criteria:

* Completed all visits in study CTBM100C2303, and visit 4 took place not more than 5 days before enrollment into this study.
* Confirmed diagnosis of cystic fibrosis participants with P. aeruginosa infection.
* Forced Expiratory Volume in One Second (FEV1) at screening (study CTBM100C2303) must be between 25% and 80% of normal predicted values.

Exclusion Criteria:

* Any use of inhaled anti-pseudomonal antibiotics between the termination of the core trial CTMB100C2303 and the enrollment into this study.
* Known local or systemic hypersensitivity to aminoglycosides or inhaled antibiotics.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2009-08-12 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Tallinn, Estonia
- Novartis Investigative Site, Yaroslavl, Russia

REFERENCES:
- [Result] Konstan MW, Flume PA, Galeva I, Wan R, Debonnett LM, Maykut RJ, Angyalosi G. One-year safety and efficacy of tobramycin powder for inhalation in patients with cystic fibrosis. Pediatr Pulmonol. 2016 Apr;51(4):372-8. doi: 10.1002/ppul.23358. Epub 2015 Dec 27. PMID 26709158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had completed all visits in the core study CTBM100C2303 took part in this extension study at 16 centers in 8 countries Bulgaria, Egypt, Estonia, Latvia, India, Lithuania, Romania and Russia from 12 August 2009 to 6 October 2011.
Pre-assignment Details: A total of 55 participants who completed all visits in the core study CTBM100C2303 and received one cycle (Cycle 1) of either Tobramycin Inhalation Powder (TIP) or matching placebo entered into the extension study and received 3 additional TIP cycles (Cycles 2, 3 and 4).
Groups:
- Tobramycin Inhalation Powder (TIP): Participants received 112 mg (four 28 mg capsules) of TIP administered by the T-326 Inhaler, twice a day (b.i.d), given in a cycle of 28 days on treatment followed by 28 days off treatment (one cycle = 56 days) for up to 3 cycles.
Period: Overall Study
Arm/Group | Tobramycin Inhalation Powder (TIP)
Started | 55
Completed | 51
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Administrative Problems | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all enrolled participants who completed their participation in the core study (CTBM100C2303) and received at least one dose of study drug in the extension study.
Groups:
- Tobramycin Inhalation Powder: Participants received 112 mg (four 28 mg capsules) of TIP administered by the T-326 Inhaler, b.i.d., given in a cycle of 28 days on treatment followed by 28 days off treatment (one cycle = 56 days) for up to 3 cycles.
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (4.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 20
Baseline Forced Expiratory Volume in One Second (FEV1) Percent Predicted [Mean (Standard Deviation); unit: percentage] — Baseline for safety analyses was defined as the last measurement prior to first drug in the core study CTBM100C2303. Population: Number analyzed were the number of participants with data available for analyses at given time point.
  percentage
    number analyzed (Participants) | 52
    (all) | 59.9 (16.24)
Baseline Forced Vital Capacity (FVC) Percent Predicted [Mean (Standard Deviation); unit: percentage] — Baseline for safety analyses was defined as the last measurement prior to first drug in the core study CTBM100C2303. Population: Number analyzed were the number of participants with data available for analyses at given time point.
  percentage
    number analyzed (Participants) | 52
    (all) | 75.2 (17.05)
Baseline Forced Expiratory Flow Rate Over 25 and 75 Percent (FEF25-75%) Predicted [Mean (Standard Deviation); unit: percentage] — Baseline for safety analyses was defined as the last measurement prior to first drug in the core study CTBM100C2303. Population: Number analyzed were the number of participants with data available for analyses at given time point.
  percentage
    number analyzed (Participants) | 52
    (all) | 37.2 (20.19)
Baseline P. aeruginosa Sputum Density [Mean (Standard Deviation); unit: log10 Colony Forming Units (CFU)] — Baseline for safety analyses was defined as the last measurement prior to first drug in the core study CTBM100C2303. Population: Number analyzed were the number of participants with data available for analyses at given time point.
  log10 Colony Forming Units (CFU)
    number analyzed (Participants) | 50
    (all) | 7.3 (1.81)
Baseline P. aeruginosa Tobramycin Minimal Inhibitory Concentration (MIC) [Mean (Standard Deviation); unit: microgram/ mL (µg/mL)] — Baseline for safety analyses was defined as the last measurement prior to first drug in the core study CTBM100C2303.
  microgram/ mL (µg/mL) | 4.6 (14.60)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal product.
Time Frame: From first administration of study drug to study completion (up to approximately 25 weeks)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage of participants | 47.3

2. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: SAEs included adverse events that resulted in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
Time Frame: From time of consent to 4 weeks after study completion (up to approximately 29 weeks)
Population: Safety Population included all enrolled participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage of participants | 5.5

3. Primary Outcome: Percentage of Death Cases
Time Frame: From time of consent to 4 weeks after study completion (up to approximately 29 weeks)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage of participants | 0

4. Primary Outcome: Percentage of Participants With Adverse Events and Serious Adverse Events Leading to Permanent Study Discontinuation
Description: AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal product. SAEs included adverse events that resulted in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
Time Frame: From first administration of study drug to study completion (up to approximately 25 weeks)
Population: Safety Population included all enrolled participants who completed their participation in the core study (CTBM100C2303) and received at least one dose of study drug in the extension study. Number analyzed were the number of participants with data available for analyses at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage of participants
  Discontinuation Due to Adverse Events | 1.8
  Discontinuation Due to Serious Adverse Events | 0

5. Primary Outcome: Shift From Baseline in Laboratory Parameters to Above Upper/Lower Limit of Normal
Description: Shift from baseline in hematology and biochemistry values to above upper/below lower limit of normal at any time post-baseline were reported. Baseline for safety analyses was defined as the last measurement prior to first dose of study drug in the core study CTBM100C2303. Change to low referred to number of participants with normal or high values at baseline. Change to high referred to number of participants with normal or low values at baseline.
Time Frame: From baseline to study completion (up to approximately 25 weeks)
Population: as for outcome 4
Measure: Number; unit: percentage of participants at risk
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage of participants at risk
  Hematology (Hem): Absolute Basophils - low: number analyzed (Participants) | 51
  Hematology (Hem): Absolute Basophils - low | 0.0
  Hem: Absolute Basophils - high: number analyzed (Participants) | 50
  Hem: Absolute Basophils - high | 16.0
  Hem: Absolute Eosinophils - low: number analyzed (Participants) | 51
  Hem: Absolute Eosinophils - low | 0.0
  Hem: Absolute Eosinophils - high: number analyzed (Participants) | 45
  Hem: Absolute Eosinophils - high | 33.3
  Hem: Absolute Lymphocytes - low: number analyzed (Participants) | 47
  Hem: Absolute Lymphocytes - low | 10.6
  Hem: Absolute Lymphocytes - high: number analyzed (Participants) | 37
  Hem: Absolute Lymphocytes - high | 32.4
  Hem: Absolute Monocytes - low: number analyzed (Participants) | 51
  Hem: Absolute Monocytes - low | 0.0
  Hem: Absolute Monocytes - high: number analyzed (Participants) | 43
  Hem: Absolute Monocytes - high | 20.9
  Hem: Absolute Neutrophils (Seg. + Bands) - low: number analyzed (Participants) | 46
  Hem: Absolute Neutrophils (Seg. + Bands) - low | 28.3
  Hem: Absolute Neutrophils (Seg. + Bands) - high: number analyzed (Participants) | 42
  Hem: Absolute Neutrophils (Seg. + Bands) - high | 35.7
  Hem: Basophils - low: number analyzed (Participants) | 51
  Hem: Basophils - low | 0.0
  Hem: Basophils - high: number analyzed (Participants) | 27
  Hem: Basophils - high | 70.4
  Hem: Eosinophils - low: number analyzed (Participants) | 51
  Hem: Eosinophils - low | 0.0
  Hem: Eosinophils - high: number analyzed (Participants) | 45
  Hem: Eosinophils - high | 37.8
  Hem: Hematocrit - low: number analyzed (Participants) | 53
  Hem: Hematocrit - low | 0.0
  Hem: Hematocrit - high: number analyzed (Participants) | 44
  Hem: Hematocrit - high | 29.5
  Hem: Hemoglobin - low: number analyzed (Participants) | 52
  Hem: Hemoglobin - low | 5.8
  Hem: Hemoglobin - high: number analyzed (Participants) | 50
  Hem: Hemoglobin - high | 6.0
  Hem: Lymphocytes - low: number analyzed (Participants) | 47
  Hem: Lymphocytes - low | 12.8
  Hem: Lymphocytes - high: number analyzed (Participants) | 43
  Hem: Lymphocytes - high | 39.5
  Hem: Monocytes - low: number analyzed (Participants) | 47
  Hem: Monocytes - low | 14.9
  Hem: Monocytes - high: number analyzed (Participants) | 40
  Hem: Monocytes - high | 42.5
  Hem: Neutrophils (Seg. + Bands) - low: number analyzed (Participants) | 45
  Hem: Neutrophils (Seg. + Bands) - low | 37.8
  Hem: Neutrophils (Seg. + Bands) - high: number analyzed (Participants) | 48
  Hem: Neutrophils (Seg. + Bands) - high | 10.4
  Hem: Platelet count (direct) - low: number analyzed (Participants) | 49
  Hem: Platelet count (direct) - low | 2.0
  Hem: Platelet count (direct) - high: number analyzed (Participants) | 25
  Hem: Platelet count (direct) - high | 24.0
  Hem: RBC- low: number analyzed (Participants) | 53
  Hem: RBC- low | 0.0
  Hem: RBC- high: number analyzed (Participants) | 36
  Hem: RBC- high | 27.8
  Hem: WBC (total)- low: number analyzed (Participants) | 44
  Hem: WBC (total)- low | 20.5
  Hem: WBC (total)- high: number analyzed (Participants) | 41
  Hem: WBC (total)- high | 31.7
  Biochemistry (Bio): Albumin - low: number analyzed (Participants) | 54
  Biochemistry (Bio): Albumin - low | 0.0
  Bio: Albumin - high: number analyzed (Participants) | 37
  Bio: Albumin - high | 32.4
  Bio: Alkaline phosphatase, serum - low: number analyzed (Participants) | 54
  Bio: Alkaline phosphatase, serum - low | 0.0
  Bio: Alkaline phosphatase, serum - high: number analyzed (Participants) | 41
  Bio: Alkaline phosphatase, serum - high | 22.0
  Bio: Bilirubin (direct/conjugated) -low: number analyzed (Participants) | 54
  Bio: Bilirubin (direct/conjugated) -low | 0.0
  Bio: Bilirubin (direct/conjugated) -high: number analyzed (Participants) | 51
  Bio: Bilirubin (direct/conjugated) -high | 11.8
  Bio: Bilirubin (total) - low | 0.0
  Bio: Bilirubin (total) - high: number analyzed (Participants) | 54
  Bio: Bilirubin (total) - high | 7.4
  Bio: Blood Urea Nitrogen (BUN) - low: number analyzed (Participants) | 48
  Bio: Blood Urea Nitrogen (BUN) - low | 16.7
  Bio: Blood Urea Nitrogen (BUN) - high | 10.9
  Bio: Calcium -low | 12.7
  Bio: Calcium - high: number analyzed (Participants) | 54
  Bio: Calcium - high | 11.1
  Bio: Chloride - low | 9.1
  Bio: Chloride - high | 1.8
  Bio: Creatinine - low: number analyzed (Participants) | 11
  Bio: Creatinine - low | 36.4
  Bio: Creatinine - high: number analyzed (Participants) | 54
  Bio: Creatinine - high | 1.9
  Bio: Gamma Glutamyltransferase - low: number analyzed (Participants) | 54
  Bio: Gamma Glutamyltransferase - low | 1.9
  Bio: Gamma Glutamyltransferase - high: number analyzed (Participants) | 48
  Bio: Gamma Glutamyltransferase - high | 10.4
  Bio: Glucose - low: number analyzed (Participants) | 50
  Bio: Glucose - low | 24.0
  Bio: Glucose - high: number analyzed (Participants) | 53
  Bio: Glucose - high | 15.1
  Bio: Phosphate (Inorganic Phosphorus) - low | 1.8
  Bio: Phosphate (Inorganic Phosphorus) - high: number analyzed (Participants) | 51
  Bio: Phosphate (Inorganic Phosphorus) - high | 47.1
  Bio: Potassium - low: number analyzed (Participants) | 53
  Bio: Potassium - low | 3.8
  Bio: Potassium - high: number analyzed (Participants) | 54
  Bio: Potassium - high | 7.4
  Bio: SGOT (AST) - low: number analyzed (Participants) | 54
  Bio: SGOT (AST) - low | 3.7
  Bio: SGOT (AST) - high: number analyzed (Participants) | 46
  Bio: SGOT (AST) - high | 30.4
  Bio: SGPT (ALT) - low: number analyzed (Participants) | 53
  Bio: SGPT (ALT) - low | 0.0
  Bio: SGPT (ALT) - high: number analyzed (Participants) | 41
  Bio: SGPT (ALT) - high | 39.0
  Bio: Serum bicarbonate - low: number analyzed (Participants) | 37
  Bio: Serum bicarbonate - low | 45.9
  Bio: Serum bicarbonate - high | 0.0
  Bio: Sodium - low | 10.9
  Bio: Sodium - high | 5.5
  Bio: Total Protein (Serum) - low | 1.8
  Bio: Total Protein (Serum) - high: number analyzed (Participants) | 43
  Bio: Total Protein (Serum) - high | 27.9
  Bio: Uric Acid - low | 1.8
  Bio: Uric Acid - high: number analyzed (Participants) | 50
  Bio: Uric Acid - high | 16.0

6. Primary Outcome: Acute Relative Change in Airways Reactivity [Forced Expiratory Value in One Second (FEV1) Percent (%) Predicted] From Pre-dose to 30 Minutes After Completion of First Dose of Study Drug
Description: Airway Reactivity was defined as ≥20% FEV1 relative decrease in percent predicted from pre dose to 30 minutes post dose. FEV1 was defined as the volume of air expired in 1 second. FEV1 % predicted was a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. Relative change in FEV1 % predicted = 100* (30 minutes post dose - pre dose) / pre dose assessed by number and percentage of participants with a decrease in ≥20% FEV1 percent predicted from pre dose to 30 minutes post dose. Baseline for was defined as the last measurement prior to first dose of study drug in the core study CTBM100C2303.
Time Frame: Pre-dose and 30 minutes Post-dose on Day 1 and Day 29 of every Cycle (2, 3, 4)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage change
  Cycle 2: Day 1: number analyzed (Participants) | 44
  Cycle 2: Day 1 | 0.0 (12.07)
  Cycle 2: Day 29: number analyzed (Participants) | 43
  Cycle 2: Day 29 | -3.0 (7.21)
  Cycle 3: Day 1: number analyzed (Participants) | 46
  Cycle 3: Day 1 | -1.4 (13.33)
  Cycle 3: Day 29: number analyzed (Participants) | 46
  Cycle 3: Day 29 | -1.8 (6.67)
  Cycle 4: Day 1: number analyzed (Participants) | 46
  Cycle 4: Day 1 | -3.0 (11.01)
  Cycle 4: Day 29: number analyzed (Participants) | 49
  Cycle 4: Day 29 | -0.6 (6.82)

7. Primary Outcome: Percentage of Participants With Frequency Decrease From Baseline in the Post-baseline Audiology Tests
Description: Auditory acuity of participants was measured using a standard dual-channel audiometer at frequencies from 250 to 8000 Hertz, and an audiogram (pure-tone air conduction) and tympanogram were performed by an audiologist. The categories reported includes >= 10dB decrease in 3 consecutive frequencies in either ear, >= 15dB decrease in 2 consecutive frequencies in either ear, and >= 20dB decrease in at least one frequency in either ear.
Time Frame: From first dose of study drug to study completion (up to approximately 25 weeks)
Population: Safety Population (Audiology Subgroup) included all participants in the safety population with at least one audiology testing. Safety Population included all enrolled participants who completed their participation in the core study (CTBM100C2303) and received at least one dose of study drug in the extension study. Number analyzed were the number of participants with normal hearing at baseline with data available for analyses at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 22
percentage of participants
  Cycle 2: Day 1; ˃= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 18
  Cycle 2: Day 1; ˃= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 5.6
  Cycle 2: Day 1: >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 18
  Cycle 2: Day 1: >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear | 0.0
  Cycle 2: Day 1; >= 20 dB Decrease in at Least One Frequency In Either Ear: number analyzed (Participants) | 18
  Cycle 2: Day 1; >= 20 dB Decrease in at Least One Frequency In Either Ear | 0.0
  Cycle 2: Day 29; ˃= 10 dB decrease in 3 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 20
  Cycle 2: Day 29; ˃= 10 dB decrease in 3 Consecutive Frequencies in Either Ear | 5.0
  Cycle 2: Day 29; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 20
  Cycle 2: Day 29; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear | 0.0
  Cycle 2: Day 29; >= 20 dB Decrease in at Least One Frequency In Either Ear: number analyzed (Participants) | 20
  Cycle 2: Day 29; >= 20 dB Decrease in at Least One Frequency In Either Ear | 0.0
  Cycle 3: Day 29; ˃= 10 dB Decrease in 3 Consecutive Frequencies in Either Ear | 9.1
  Cycle 3: Day 29; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear | 4.5
  Cycle 3: Day 29; >= 20 dB Decrease in at Least One Frequency In Either Ear | 4.5
  Cycle 4: Day 29; ˃= 10 dB decrease in 3 Consecutive Frequencies in Either Ear | 4.5
  Cycle 4: Day 29; >= 15 dB Decrease In 2 Consecutive Frequencies in Either Ear | 0.0
  Cycle 4: Day 29; >= 20 dB Decrease in at Least One Frequency In Either Ear | 0.0
  Follow Up: Day 57; ˃= 10 dB decrease in 3 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 8
  Follow Up: Day 57; ˃= 10 dB decrease in 3 Consecutive Frequencies in Either Ear | 0.0
  Follow Up: Day 57: >= 15 dB Decrease in 2 Consecutive Frequencies in Either Ear: number analyzed (Participants) | 8
  Follow Up: Day 57: >= 15 dB Decrease in 2 Consecutive Frequencies in Either Ear | 0.0
  Follow Up: Day 57; >= 20 dB Decrease in at Least One Frequency In Either Ear: number analyzed (Participants) | 8
  Follow Up: Day 57; >= 20 dB Decrease in at Least One Frequency In Either Ear | 0.0

8. Primary Outcome: Number of Participants With Adverse Events (AEs) Associated With the Use of New Antipseudomonal Antibiotic
Description: as for outcome 4
Time Frame: From first administration of study drug to study completion (up to approximately 25 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
Participants
  Mild, Yes | 1
  Mild, No | 13
  Moderate, Yes | 3
  Moderate, No | 9
  Severe, Yes | 0
  Severe, No | 0

9. Secondary Outcome: Relative Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Percent Predicted to End of Dosing at Each Cycle and Study Completion
Description: FEV1 was defined as the volume of air expired in 1 second. FEV1 % predicted was a normalized value of FEV1 calculated using the Knudsen equation, based upon participant's age, gender and height. Relative change in FEV1 % predicted = 100* (30 minutes post dose - pre dose) / pre dose assessed by number and percentage of participants with a decrease in ≥20% FEV1 percent predicted from pre dose to 30 minutes post dose. Baseline for was defined as the last measurement prior to first dose of study drug in the core study CTBM100C2303. Termination referred to the last available pre dose post-baseline measurement.
Time Frame: Baseline, Day 29 of Cycle 2, 3, 4, Day 57 of Follow Up and Termination (Study Completion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage change
  Cycle 2: Day 29: number analyzed (Participants) | 47
  Cycle 2: Day 29 | 13.5 (23.42)
  Cycle 3: Day 29: number analyzed (Participants) | 49
  Cycle 3: Day 29 | 14.8 (22.40)
  Cycle 4: Day 29: number analyzed (Participants) | 48
  Cycle 4: Day 29 | 17.3 (23.56)
  Follow Up: Day 57: number analyzed (Participants) | 47
  Follow Up: Day 57 | 13.5 (20.62)
  Termination: number analyzed (Participants) | 52
  Termination | 13.9 (21.86)

10. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) Percent (%) Predicted to End of Dosing at Each Cycle and Study Completion
Description: Relative change from baseline in FVC % predicted to end of dosing in each cycle and study completion were reported. Relative change from baseline was defined as: Relative change = 100* (Post baseline- baseline) / baseline. Baseline was defined as last measurement prior to first dose of study drug in the core study CTBM100C2303. Termination referred to the last available pre dose post-baseline measurement.
Time Frame: Baseline, Day 29 of Cycle 2, 3, 4, Day 57 of Follow Up and Termination (Study Completion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage change
  Cycle 2: Day 29: number analyzed (Participants) | 47
  Cycle 2: Day 29 | 7.0 (17.46)
  Cycle 3: Day 29: number analyzed (Participants) | 49
  Cycle 3: Day 29 | 7.2 (16.89)
  Cycle 4: Day 29: number analyzed (Participants) | 48
  Cycle 4: Day 29 | 9.6 (16.87)
  Follow Up: Day 57: number analyzed (Participants) | 47
  Follow Up: Day 57 | 7.4 (14.99)
  Termination: number analyzed (Participants) | 52
  Termination | 7.9 (15.24)

11. Secondary Outcome: Change From Baseline in Forced Expiratory Flow Rate Over 25 Percent and 75 Percent (FEF25-75%) Predicted to End of Dosing at Each Cycle and Study Completion
Description: Relative change from baseline in FEF25-75% predicted to end of dosing in each cycle and study completion were reported. Relative change from baseline was defined as: Relative change = 100* (Post baseline- baseline) / baseline. Baseline was defined as last measurement prior to first dose of study drug in the core study CTBM100C2303. Termination referred to the last available pre dose post-baseline measurement.
Time Frame: Baseline, Day 29 of Cycle 2, 3, 4, Day 57 of Follow Up and Termination (Study Completion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage change
  Cycle 2: Day 29: number analyzed (Participants) | 47
  Cycle 2: Day 29 | 35.2 (55.86)
  Cycle 3: Day 29: number analyzed (Participants) | 49
  Cycle 3: Day 29 | 44.7 (58.17)
  Cycle 4; Day 29: number analyzed (Participants) | 48
  Cycle 4; Day 29 | 40.5 (59.21)
  Follow Up: Day 57: number analyzed (Participants) | 47
  Follow Up: Day 57 | 35.9 (58.08)
  Termination: number analyzed (Participants) | 52
  Termination | 34.7 (57.98)

12. Secondary Outcome: Absolute Change From Baseline in Sputum Pseudomonas Aeruginosa Density [log10 Colony Forming Units (CFU) Per Gram Sputum] to End of Dosing at Each Cycle and Study Completion
Description: P. aeruginosa sputum density referred to overall density, defined as the sum of biotypes (mucoid, dry and small colony variant). If sub-isolates existed for CFU biotype mucoid or dry, then the sum of sub-isolates was analyzed. Absolute change from baseline was defined as: Absolute change = Post Baseline - Baseline. Baseline was defined as last measurement prior to first dose of study drug in the core study CTBM100C2303. Termination referred to the last available pre dose post-baseline measurement.
Time Frame: Baseline, Day 29 of Cycle 2, 3, 4, Day 57 of Follow Up and Termination (Study Completion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 Colony Forming Units (CFU)
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
log10 Colony Forming Units (CFU)
  Cycle 2: Day 29: number analyzed (Participants) | 46
  Cycle 2: Day 29 | -3.7 (2.76)
  Cycle 3: Day 29: number analyzed (Participants) | 49
  Cycle 3: Day 29 | -3.5 (3.04)
  Cycle 4: Day 29: number analyzed (Participants) | 44
  Cycle 4: Day 29 | -3.9 (2.82)
  Follow Up: Day 57: number analyzed (Participants) | 23
  Follow Up: Day 57 | -1.1 (2.82)
  Termination: number analyzed (Participants) | 50
  Termination | -2.9 (3.16)

13. Secondary Outcome: Change From Baseline in Pseudomonas Aeruginosa Minimum Inhibitory Concentration (MIC) to End of Dosing at Each Cycle and Study Completion
Description: Change in tobramycin MIC values for P. aeruginosa were reported for specimens and were used to assess the change in pathogen susceptibility to tobramycin before (baseline) and after (post-baseline) the treatment. Maximum MIC values from all biotypes were used. Change from baseline was defined as: Change = Post-baseline - Baseline. Baseline was defined as last measurement prior to first dose of study drug in the core studyCTBM100C2303.Termination referred to the last available pre dose post-baseline measurement.
Time Frame: Baseline, Day 29 of Cycle 2, 3, 4, Day 57 of Follow Up and Termination (Study Completion)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
μg/mL
  Cycle 2: Day 29: number analyzed (Participants) | 39
  Cycle 2: Day 29 | 15.1 (82.45)
  Cycle 3: Day 29: number analyzed (Participants) | 41
  Cycle 3: Day 29 | 30.7 (112.32)
  Cycle 4: Day 29: number analyzed (Participants) | 35
  Cycle 4: Day 29 | 24.0 (90.13)
  Follow Up: Day 57: number analyzed (Participants) | 21
  Follow Up: Day 57 | 28.6 (111.71)
  Termination: number analyzed (Participants) | 51
  Termination | 22.3 (101.38)

14. Secondary Outcome: Percentage of Participants With Anti-Pseudomonal Antibiotic Use During The Treatment Period
Time Frame: From first administration of study drug to study completion (up to approximately 25 weeks)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
percentage of participants | 9.1

15. Secondary Outcome: Number of Days of Hospitalization Due to Respiratory Serious Adverse Events
Description: SAEs included adverse events that resulted in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. For calculation of days in hospitalization due to respiratory events, the end date was defined as the discharge date (if provided and even if after the end of the extension study), and otherwise as the date of last visit.
Time Frame: From first administration of study drug to study completion (up to approximately 25 weeks)
Population: as for baseline characteristics
Measure: Median (Full Range); unit: days
Arm/Group | Tobramycin Inhalation Powder
Number analyzed (Participants) | 55
days | 13.0 [8.0 to 18.0]

ADVERSE EVENTS:
Time Frame: From first administration of study drug to study completion (up to approximately 25 weeks)
Description: Safety Population included all enrolled participants who completed their participation in the core study (CTBM100C2303) and received at least one dose of study drug in the extension study.
Arm/Group | Tobramycin Inhalation Powder
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 3/55
Other Adverse Events (participants affected / at risk) | 24/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (N=55)
Aspergillosis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tobramycin Inhalation Powder (N=55)
Hypoacusis (Ear and labyrinth disorders) | 3
Middle ear effusion (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 2
Ascariasis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2
Gastrointestinal candidiasis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 5
Respiratory tract infection viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Stenotrophomonas infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral rhinitis (Infections and infestations) | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1
Blood calcium decreased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Protein urine (Investigations) | 1
Protein urine present (Investigations) | 2
White blood cell count increased (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.